CLINICAL TRIAL: NCT01078584
Title: A Prospective, Non-interventional, Observational Study To Describe the Effectiveness of Trandolapril (Mavik®) in the Management of Patients Requiring Angiotensin Converting Enzyme Inhibitor Treatment (In-MAU-tion)
Brief Title: Canadian Study of Trandolapril on Blood Pressure in Hypertensive Patients
Acronym: in-MAU-tion
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Collaborators: McKesson Canada (Network)
Responsible Party: Sponsor
Other Study IDs: P10-665
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Results first posted 2012-10-11 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Hypertension
Keywords: Uncontrolled hypertension; trandolapril
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Hypertensive Participants: Hypertensive diabetics and non-diabetics, with or without isolated systemic hypertension and/or renal dysfunction, who were naïve to trandolapril or on trandolapril within past 30 days.

SUMMARY:
The in-MAU-tion study is conducted to determine the percentage of hypertensive participants with or without diabetes reaching CHEP (Canadian Hypertension Education Program) defined blood pressure targets. Additionally, the study assesses change in renal function (microalbuminuria, estimated glomerular filtration rate) in hypertensive participants treated with trandolapril (Mavik®) and examines patient satisfaction with trandolapril (Mavik®) therapy.

DETAILED DESCRIPTION:
There are no interventional implications in this study. The study runs under consideration of Canadian Hypertension Education Program guidelines and as per standard practice of care. Data collection is recorded on the appropriate case report forms. The data collected consist of: patient demographics (gender, race, age, weight), blood pressure readings, heart rate, coexisting comorbidities, concomitant chronic medications (generic name and dosage), indication and dose for trandolapril (Mavik®) and patient compliance. Laboratory values (microalbuminuria, estimated glomerular filtration rate) are only collected if the data are available for each patient. For baseline values (study Day 0), any laboratory value recorded within the past year prior to the baseline visit (Visit 1) is recorded, if the value is available. As per Canadian Hypertension Education Program recommendations and as a support and educational measure, patients are provided with (1) educational tools (nutrition guidebooks) and (2) home blood pressure monitoring devices. As per research and development guidelines, blood pressure devices were retrieved at the end of the study. Approximately 8,000 hypertensive participants were enrolled in the study at up to 700 sites across Canada. Sample size estimations were based on the assumption that 67.2% of non-diabetic hypertensive participants (assumed to make up to 69% of the eligible participant population) would reach a blood pressure target of <140/90mm Hg, while 22% of diabetes participants (31% of the eligible population) would meet a blood pressure target of <130/80 mm Hg with trandolapril (Mavik®) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults capable of providing consent and who have uncontrolled hypertension
* Participants were either treatment-naïve or had uncontrolled hypertension on their existing antihypertensive medication.

Exclusion Criteria:

* Participants were excluded from participation in the study if they had been taking trandolapril (Mavik®), alone or in combination, for more than 1 month prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 7993 (Actual)
Dates: Start 2008-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Assouline, PhD, Study Director — Abbott
Locations (568):
- Canada (568):
  - Site Reference ID/Investigator# 32207, Calgary, Alberta
  - Site Reference ID/Investigator# 10283, Calgary, Alberta
  - Site Reference ID/Investigator# 32168, Calgary, Alberta
  - Site Reference ID/Investigator# 32147, Calgary, Alberta
  - Site Reference ID/Investigator# 42438, Calgary, Alberta
  - Site Reference ID/Investigator# 32157, Calgary, Alberta
  - Site Reference ID/Investigator# 37940, Calgary, Alberta
  - Site Reference ID/Investigator# 32199, Calgary, Alberta
  - Site Reference ID/Investigator# 32144, Calgary, Alberta
  - Site Reference ID/Investigator# 32169, Calgary, Alberta
  - Site Reference ID/Investigator# 42391, Edmonton, Alberta
  - Site Reference ID/Investigator# 32146, Edmonton, Alberta
  - Site Reference ID/Investigator# 32165, Edmonton, Alberta
  - Site Reference ID/Investigator# 32197, Edmonton, Alberta
  - Site Reference ID/Investigator# 32126, Edmonton, Alberta
  - Site Reference ID/Investigator# 37892, Edmonton, Alberta
  - Site Reference ID/Investigator# 32178, Edmonton, Alberta
  - Site Reference ID/Investigator# 42406, Edmonton, Alberta
  - Site Reference ID/Investigator# 32160, Edmonton, Alberta
  - Site Reference ID/Investigator# 32200, Edmonton, Alberta
  - Site Reference ID/Investigator# 32149, Edmonton, Alberta
  - Site Reference ID/Investigator# 32156, Edmonton, Alberta
  - Site Reference ID/Investigator# 32216, Edmonton, Alberta
  - Site Reference ID/Investigator# 32206, Edmonton, Alberta
  - Site Reference ID/Investigator# 32128, Red Deer, Alberta
  - Site Reference ID/Investigator# 32175, Red Deer, Alberta
  - Site Reference ID/Investigator# 32124, Spruce Grove, Alberta
  - Site Reference ID/Investigator# 37846, 100 Mile House, British Columbia
  - Site Reference ID/Investigator# 30893, Abbotsford, British Columbia
  - Site Reference ID/Investigator# 37728, Abbotsford, British Columbia
  - Site Reference ID/Investigator# 31375, Aldergrove, British Columbia
  - Site Reference ID/Investigator# 30870, Burnaby, British Columbia
  - Site Reference ID/Investigator# 30964, Burnaby, British Columbia
  - Site Reference ID/Investigator# 31261, Burnaby, British Columbia
  - Site Reference ID/Investigator# 30946, Burnaby, British Columbia
  - Site Reference ID/Investigator# 30927, Burnaby, British Columbia
  - Site Reference ID/Investigator# 42433, Coquitlam, British Columbia
  - Site Reference ID/Investigator# 32213, Coquitlam, British Columbia
  - Site Reference ID/Investigator# 32166, Delta, British Columbia
  - Site Reference ID/Investigator# 31288, Delta, British Columbia
  - Site Reference ID/Investigator# 42404, Delta, British Columbia
  - Site Reference ID/Investigator# 37922, Delta, British Columbia
  - Site Reference ID/Investigator# 30926, Delta, British Columbia
  - Site Reference ID/Investigator# 37666, Kamloops, British Columbia
  - Site Reference ID/Investigator# 30929, Kamloops, British Columbia
  - Site Reference ID/Investigator# 32203, Kamloops, British Columbia
  - Site Reference ID/Investigator# 37882, Kamloops, British Columbia
  - Site Reference ID/Investigator# 42365, Kelowna, British Columbia
  - Site Reference ID/Investigator# 33018, Kelowna, British Columbia
  - Site Reference ID/Investigator# 30915, Kelowna, British Columbia
  - Site Reference ID/Investigator# 33043, Langley, British Columbia
  - Site Reference ID/Investigator# 31315, Maple Ridge, British Columbia
  - Site Reference ID/Investigator# 33234, North Vancouver, British Columbia
  - Site Reference ID/Investigator# 32433, Penticton, British Columbia
  - Site Reference ID/Investigator# 32435, Pitt Meadows, British Columbia
  - Site Reference ID/Investigator# 30884, Port Coquitlam, British Columbia
  - Site Reference ID/Investigator# 32467, Richmond, British Columbia
  - Site Reference ID/Investigator# 37671, Richmond, British Columbia
  - Site Reference ID/Investigator# 30890, Surrey, British Columbia
  - Site Reference ID/Investigator# 31278, Surrey, British Columbia
  - Site Reference ID/Investigator# 37888, Surrey, British Columbia
  - Site Reference ID/Investigator# 30966, Surrey, British Columbia
  - Site Reference ID/Investigator# 42332, Surrey, British Columbia
  - Site Reference ID/Investigator# 37780, Surrey, British Columbia
  - Site Reference ID/Investigator# 31383, Surrey, British Columbia
  - Site Reference ID/Investigator# 42422, Surrey, British Columbia
  - Site Reference ID/Investigator# 30867, Trail, British Columbia
  - Site Reference ID/Investigator# 30916, Trail, British Columbia
  - Site Reference ID/Investigator# 30908, Vancouver, British Columbia
  - Site Reference ID/Investigator# 33122, Vancouver, British Columbia
  - Site Reference ID/Investigator# 31396, Vancouver, British Columbia
  - Site Reference ID/Investigator# 30919, Vancouver, British Columbia
  - Site Reference ID/Investigator# 37725, Vancouver, British Columbia
  - Site Reference ID/Investigator# 33123, Vancouver, British Columbia
  - Site Reference ID/Investigator# 37771, Vancouver, British Columbia
  - Site Reference ID/Investigator# 31316, Victoria, British Columbia
  - Site Reference ID/Investigator# 31277, Victoria, British Columbia
  - Site Reference ID/Investigator# 32177, Victoria, British Columbia
  - Site Reference ID/Investigator# 33128, Victoria, British Columbia
  - Site Reference ID/Investigator# 33129, Victoria, British Columbia
  - Site Reference ID/Investigator# 30938, Victoria, British Columbia
  - Site Reference ID/Investigator# 32120, Victoria, British Columbia
  - Site Reference ID/Investigator# 30952, Victoria, British Columbia
  - Site Reference ID/Investigator# 31320, Victoria, British Columbia
  - Site Reference ID/Investigator# 32191, West Vancouver, British Columbia
  - Site Reference ID/Investigator# 30951, Whitby, British Columbia
  - Site Reference ID/Investigator# 32227, Brandon, Manitoba
  - Site Reference ID/Investigator# 30933, Gimli, Manitoba
  - Site Reference ID/Investigator# 31328, Stonewall, Manitoba
  - Site Reference ID/Investigator# 31376, Stonewall, Manitoba
  - Site Reference ID/Investigator# 31306, Winnipeg, Manitoba
  - Site Reference ID/Investigator# 31395, Winnipeg, Manitoba
  - Site Reference ID/Investigator# 33169, Winnipeg, Manitoba
  - Site Reference ID/Investigator# 33167, Winnipeg, Manitoba
  - Site Reference ID/Investigator# 32180, Winnipeg, Manitoba
  - Site Reference ID/Investigator# 30901, Winnipeg, Manitoba
  - Site Reference ID/Investigator# 33173, Winnipeg, Manitoba
  - Site Reference ID/Investigator# 33171, Winnipeg, Manitoba
  - Site Reference ID/Investigator# 32122, Winnipeg, Manitoba
  - Site Reference ID/Investigator# 33172, Winnipeg, Manitoba
  - Site Reference ID/Investigator# 33174, Winnipeg, Manitoba
  - Site Reference ID/Investigator# 33166, Winnipeg, Manitoba
  - Site Reference ID/Investigator# 31263, Winnipeg, Manitoba
  - Site Reference ID/Investigator# 32209, Dieppe, New Brunswick
  - Site Reference ID/Investigator# 32212, Moncton, New Brunswick
  - Site Reference ID/Investigator# 32211, Saint-Louis de Kent, New Brunswick
  - Site Reference ID/Investigator# 31322, Sussex, New Brunswick
  - Site Reference ID/Investigator# 30878, Conception Bay South, Newfoundland and Labrador
  - Site Reference ID/Investigator# 30957, Marystown, Newfoundland and Labrador
  - Site Reference ID/Investigator# 33094, Marystown, Newfoundland and Labrador
  - Site Reference ID/Investigator# 32154, Mount Pearl, Newfoundland and Labrador
  - Site Reference ID/Investigator# 33193, Mount Pearl, Newfoundland and Labrador
  - Site Reference ID/Investigator# 30892, St. John's, Newfoundland and Labrador
  - Site Reference ID/Investigator# 30936, St. John's, Newfoundland and Labrador
  - Site Reference ID/Investigator# 31314, Bridgewater, Nova Scotia
  - Site Reference ID/Investigator# 31276, Bridgewater, Nova Scotia
  - Site Reference ID/Investigator# 31264, Dartmouth, Nova Scotia
  - Site Reference ID/Investigator# 31321, Dartmouth, Nova Scotia
  - Site Reference ID/Investigator# 31327, Halifax, Nova Scotia
  - Site Reference ID/Investigator# 37781, Kentville, Nova Scotia
  - Site Reference ID/Investigator# 33072, Lower Sackville, Nova Scotia
  - Site Reference ID/Investigator# 30894, Lower Sackville, Nova Scotia
  - Site Reference ID/Investigator# 42461, Middleton, Nova Scotia
  - Site Reference ID/Investigator# 32508, Sheet Harbour, Nova Scotia
  - Site Reference ID/Investigator# 31352, Shubencadie, Nova Scotia
  - Site Reference ID/Investigator# 42403, Truro, Nova Scotia
  - Site Reference ID/Investigator# 33165, Windsor, Nova Scotia
  - Site Reference ID/Investigator# 42367, Ajax, Ontario
  - Site Reference ID/Investigator# 42464, Ameherstburg, Ontario
  - Site Reference ID/Investigator# 37885, Amherstview, Ontario
  - Site Reference ID/Investigator# 42409, Aurora, Ontario
  - Site Reference ID/Investigator# 42449, Aurora, Ontario
  - Site Reference ID/Investigator# 30943, Aurora, Ontario
  - Site Reference ID/Investigator# 30963, Barrie, Ontario
  - Site Reference ID/Investigator# 30954, Belleville, Ontario
  - Site Reference ID/Investigator# 30879, Belleville, Ontario
  - Site Reference ID/Investigator# 42378, Bolton, Ontario
  - Site Reference ID/Investigator# 30888, Bowmanville, Ontario
  - Site Reference ID/Investigator# 30947, Bowmanville, Ontario
  - Site Reference ID/Investigator# 31286, Bradford, Ontario
  - Site Reference ID/Investigator# 32192, Bradford, Ontario
  - Site Reference ID/Investigator# 37911, Brampton, Ontario
  - Site Reference ID/Investigator# 37932, Brampton, Ontario
  - Site Reference ID/Investigator# 30882, Brampton, Ontario
  - Site Reference ID/Investigator# 37929, Brampton, Ontario
  - Site Reference ID/Investigator# 37768, Brantford, Ontario
  - Site Reference ID/Investigator# 37934, Burlington, Ontario
  - Site Reference ID/Investigator# 32173, Burlington, Ontario
  - Site Reference ID/Investigator# 32210, Burlington, Ontario
  - Site Reference ID/Investigator# 37919, Burlington, Ontario
  - Site Reference ID/Investigator# 31359, Burlington, Ontario
  - Site Reference ID/Investigator# 37923, Burlington, Ontario
  - Site Reference ID/Investigator# 37845, Burlington, Ontario
  - Site Reference ID/Investigator# 47571, Collingwood, Ontario
  - Site Reference ID/Investigator# 30956, Cornwall, Ontario
  - Site Reference ID/Investigator# 30969, Corunna, Ontario
  - Site Reference ID/Investigator# 30961, Dashwood, Ontario
  - Site Reference ID/Investigator# 37850, Dolbeau-Mistassini, Ontario
  - Site Reference ID/Investigator# 42389, Durham, Ontario
  - Site Reference ID/Investigator# 42385, East York, Ontario
  - Site Reference ID/Investigator# 42397, East York, Ontario
  - Site Reference ID/Investigator# 42400, East York, Ontario
  - Site Reference ID/Investigator# 42423, East York, Ontario
  - Site Reference ID/Investigator# 30930, East York, Ontario
  - Site Reference ID/Investigator# 31363, East York, Ontario
  - Site Reference ID/Investigator# 42342, Elmvale, Ontario
  - Site Reference ID/Investigator# 32873, Etobicoke, Ontario
  - Site Reference ID/Investigator# 31353, Etobicoke, Ontario
  - Site Reference ID/Investigator# 37774, Etobicoke, Ontario
  - Site Reference ID/Investigator# 32871, Etobicoke, Ontario
  - Site Reference ID/Investigator# 32870, Etobicoke, Ontario
  - Site Reference ID/Investigator# 32872, Etobicoke, Ontario
  - Site Reference ID/Investigator# 32880, Fonthill, Ontario
  - Site Reference ID/Investigator# 30873, Fort Erie, Ontario
  - Site Reference ID/Investigator# 31310, Fort Erie, Ontario
  - Site Reference ID/Investigator# 31356, Fort Erie, Ontario
  - Site Reference ID/Investigator# 31367, Georgetown, Ontario
  - Site Reference ID/Investigator# 31381, Georgetown, Ontario
  - Site Reference ID/Investigator# 37672, Greater Sudbury, Ontario
  - Site Reference ID/Investigator# 37674, Greater Sudbury, Ontario
  - Site Reference ID/Investigator# 31271, Greater Sudbury, Ontario
  - Site Reference ID/Investigator# 37784, Greater Sudbury, Ontario
  - Site Reference ID/Investigator# 32529, Greater Sudbury, Ontario
  - Site Reference ID/Investigator# 30965, Grimsby, Ontario
  - Site Reference ID/Investigator# 31285, Grimsby, Ontario
  - Site Reference ID/Investigator# 42347, Guelph, Ontario
  - Site Reference ID/Investigator# 42462, Guelph, Ontario
  - Site Reference ID/Investigator# 31282, Hamilton, Ontario
  - Site Reference ID/Investigator# 32223, Hamilton, Ontario
  - Site Reference ID/Investigator# 42440, Hamilton, Ontario
  - Site Reference ID/Investigator# 32214, Hamilton, Ontario
  - Site Reference ID/Investigator# 30924, Hamilton, Ontario
  - Site Reference ID/Investigator# 31348, Hamilton, Ontario
  - Site Reference ID/Investigator# 30940, Hamilton, Ontario
  - Site Reference ID/Investigator# 37907, Hamilton, Ontario
  - Site Reference ID/Investigator# 31389, Hamilton, Ontario
  - Site Reference ID/Investigator# 31275, Hamilton, Ontario
  - Site Reference ID/Investigator# 32965, Hawkesbury, Ontario
  - Site Reference ID/Investigator# 31373, Hawkesbury, Ontario
  - Site Reference ID/Investigator# 33002, Jarvis, Ontario
  - Site Reference ID/Investigator# 30876, Jordan Station, Ontario
  - Site Reference ID/Investigator# 32611, Keswick, Ontario
  - Site Reference ID/Investigator# 33020, Keswick, Ontario
  - Site Reference ID/Investigator# 31386, Kirkfield, Ontario
  - Site Reference ID/Investigator# 42443, Kitchener, Ontario
  - Site Reference ID/Investigator# 30895, Kitchener, Ontario
  - Site Reference ID/Investigator# 37783, Kitchener, Ontario
  - Site Reference ID/Investigator# 37906, Kitchener, Ontario
  - Site Reference ID/Investigator# 42467, Kitchener, Ontario
  - Site Reference ID/Investigator# 32174, La Salle, Ontario
  - Site Reference ID/Investigator# 37910, La Salle, Ontario
  - Site Reference ID/Investigator# 31347, LaSalle, Ontario
  - Site Reference ID/Investigator# 32220, Lindsay, Ontario
  - Site Reference ID/Investigator# 42348, Lindsay, Ontario
  - Site Reference ID/Investigator# 32196, London, Ontario
  - Site Reference ID/Investigator# 30900, London, Ontario
  - Site Reference ID/Investigator# 33070, London, Ontario
  - Site Reference ID/Investigator# 31333, London, Ontario
  - Site Reference ID/Investigator# 32148, London, Ontario
  - Site Reference ID/Investigator# 31340, London, Ontario
  - Site Reference ID/Investigator# 31385, Markham, Ontario
  - Site Reference ID/Investigator# 33091, Markham, Ontario
  - Site Reference ID/Investigator# 33090, Markham, Ontario
  - Site Reference ID/Investigator# 42337, Markham, Ontario
  - Site Reference ID/Investigator# 30967, Milton, Ontario
  - Site Reference ID/Investigator# 33104, Mississauga, Ontario
  - Site Reference ID/Investigator# 42398, Mississauga, Ontario
  - Site Reference ID/Investigator# 33106, Mississauga, Ontario
  - Site Reference ID/Investigator# 30945, Mississauga, Ontario
  - Site Reference ID/Investigator# 33105, Mississauga, Ontario
  - Site Reference ID/Investigator# 37673, Mississauga, Ontario
  - Site Reference ID/Investigator# 42331, Mississauga, Ontario
  - Site Reference ID/Investigator# 42373, Mississauga, Ontario
  - Site Reference ID/Investigator# 42468, Mississauga, Ontario
  - Site Reference ID/Investigator# 32152, Mississauga, Ontario
  - Site Reference ID/Investigator# 37723, Mississauga, Ontario
  - Site Reference ID/Investigator# 37903, Mississauga, Ontario
  - Site Reference ID/Investigator# 37904, Mississauga, Ontario
  - Site Reference ID/Investigator# 31312, Mississauga, Ontario
  - Site Reference ID/Investigator# 42327, Nepean, Ontario
  - Site Reference ID/Investigator# 31364, Nepean, Ontario
  - Site Reference ID/Investigator# 31334, Nepean, Ontario
  - Site Reference ID/Investigator# 31357, Newboro, Ontario
  - Site Reference ID/Investigator# 42445, Newcastle, Ontario
  - Site Reference ID/Investigator# 37770, Newmarket, Ontario
  - Site Reference ID/Investigator# 30970, Newmarket, Ontario
  - Site Reference ID/Investigator# 31388, Newmarket, Ontario
  - Site Reference ID/Investigator# 37930, Newmarket, Ontario
  - Site Reference ID/Investigator# 32172, Niagara Falls, Ontario
  - Site Reference ID/Investigator# 31326, North Bay, Ontario
  - Site Reference ID/Investigator# 30913, North Bay, Ontario
  - Site Reference ID/Investigator# 30937, North York, Ontario
  - Site Reference ID/Investigator# 32601, North York, Ontario
  - Site Reference ID/Investigator# 32602, North York, Ontario
  - Site Reference ID/Investigator# 42442, North York, Ontario
  - Site Reference ID/Investigator# 30896, North York, Ontario
  - Site Reference ID/Investigator# 31265, North York, Ontario
  - Site Reference ID/Investigator# 32607, North York, Ontario
  - Site Reference ID/Investigator# 42407, North York, Ontario
  - Site Reference ID/Investigator# 42435, North York, Ontario
  - Site Reference ID/Investigator# 33235, North York, Ontario
  - Site Reference ID/Investigator# 31350, Oakville, Ontario
  - Site Reference ID/Investigator# 37842, Oakville, Ontario
  - Site Reference ID/Investigator# 30910, Oshawa, Ontario
  - Site Reference ID/Investigator# 30971, Oshawa, Ontario
  - Site Reference ID/Investigator# 42459, Oshawa, Ontario
  - Site Reference ID/Investigator# 42415, Oshawa, Ontario
  - Site Reference ID/Investigator# 32162, Oshawa, Ontario
  - Site Reference ID/Investigator# 33260, Oshawa, Ontario
  - Site Reference ID/Investigator# 42363, Oshawa, Ontario
  - Site Reference ID/Investigator# 32164, Oshawa, Ontario
  - Site Reference ID/Investigator# 32185, Ottawa, Ontario
  - Site Reference ID/Investigator# 37884, Ottawa, Ontario
  - Site Reference ID/Investigator# 32422, Ottawa, Ontario
  - Site Reference ID/Investigator# 33267, Ottawa, Ontario
  - Site Reference ID/Investigator# 42425, Ottawa, Ontario
  - Site Reference ID/Investigator# 32190, Ottawa, Ontario
  - Site Reference ID/Investigator# 31380, Ottawa, Ontario
  - Site Reference ID/Investigator# 31287, Ottawa, Ontario
  - Site Reference ID/Investigator# 33266, Ottawa, Ontario
  - Site Reference ID/Investigator# 31301, Ottawa, Ontario
  - Site Reference ID/Investigator# 37785, Owen Sound, Ontario
  - Site Reference ID/Investigator# 42351, Pickering, Ontario
  - Site Reference ID/Investigator# 42417, Pickering, Ontario
  - Site Reference ID/Investigator# 42418, Pickering, Ontario
  - Site Reference ID/Investigator# 42419, Pickering, Ontario
  - Site Reference ID/Investigator# 37848, Pickering, Ontario
  - Site Reference ID/Investigator# 42434, Pickering, Ontario
  - Site Reference ID/Investigator# 32466, Richmond, Ontario
  - Site Reference ID/Investigator# 32468, Richmond, Ontario
  - Site Reference ID/Investigator# 32184, Richmond Hill, Ontario
  - Site Reference ID/Investigator# 32224, Richmond Hill, Ontario
  - Site Reference ID/Investigator# 30932, Richmond Hill, Ontario
  - Site Reference ID/Investigator# 31270, Richmond Hill, Ontario
  - Site Reference ID/Investigator# 30872, Richmond Hill, Ontario
  - Site Reference ID/Investigator# 37668, Saint Catherines, Ontario
  - Site Reference ID/Investigator# 32171, Saint Catherines, Ontario
  - Site Reference ID/Investigator# 37664, Sarnia, Ontario
  - Site Reference ID/Investigator# 37759, Sault Ste. Marie, Ontario
  - Site Reference ID/Investigator# 37772, Sault Ste. Marie, Ontario
  - Site Reference ID/Investigator# 42469, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 37895, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 42457, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 30942, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 37739, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 30912, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 32495, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 42421, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 42441, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 31346, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 37890, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 30906, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 42439, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 31305, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 42410, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 30958, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 42369, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 30939, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 30960, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 31382, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 47576, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 37916, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 31296, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 32494, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 42408, Scarborough Village, Ontario
  - Site Reference ID/Investigator# 32219, Schomberg, Ontario
  - Site Reference ID/Investigator# 42325, Smiths Falls, Ontario
  - Site Reference ID/Investigator# 31365, Smiths Falls, Ontario
  - Site Reference ID/Investigator# 32514, Southampton, Ontario
  - Site Reference ID/Investigator# 37777, St. Catharines, Ontario
  - Site Reference ID/Investigator# 32201, Stirling, Ontario
  - Site Reference ID/Investigator# 42387, Stirling, Ontario
  - Site Reference ID/Investigator# 42333, Stoney Creek, Ontario
  - Site Reference ID/Investigator# 32181, Stoney Creek, Ontario
  - Site Reference ID/Investigator# 37889, Surrey, Ontario
  - Site Reference ID/Investigator# 37662, Tecumseh, Ontario
  - Site Reference ID/Investigator# 37663, Tecumseh, Ontario
  - Site Reference ID/Investigator# 42392, Thornbury, Ontario
  - Site Reference ID/Investigator# 32536, Thornhill, Ontario
  - Site Reference ID/Investigator# 31300, Thunder Bay, Ontario
  - Site Reference ID/Investigator# 37938, Thunder Bay, Ontario
  - Site Reference ID/Investigator# 37787, Timmins, Ontario
  - Site Reference ID/Investigator# 37913, Timmins, Ontario
  - Site Reference ID/Investigator# 32539, Toronto, Ontario
  - Site Reference ID/Investigator# 32548, Toronto, Ontario
  - Site Reference ID/Investigator# 33044, Toronto, Ontario
  - Site Reference ID/Investigator# 42350, Toronto, Ontario
  - Site Reference ID/Investigator# 42446, Toronto, Ontario
  - Site Reference ID/Investigator# 32544, Toronto, Ontario
  - Site Reference ID/Investigator# 30920, Toronto, Ontario
  - Site Reference ID/Investigator# 32546, Toronto, Ontario
  - Site Reference ID/Investigator# 42381, Toronto, Ontario
  - Site Reference ID/Investigator# 32121, Toronto, Ontario
  - Site Reference ID/Investigator# 31269, Toronto, Ontario
  - Site Reference ID/Investigator# 30925, Toronto, Ontario
  - Site Reference ID/Investigator# 37853, Toronto, Ontario
  - Site Reference ID/Investigator# 31354, Toronto, Ontario
  - Site Reference ID/Investigator# 32542, Toronto, Ontario
  - Site Reference ID/Investigator# 37931, Toronto, Ontario
  - Site Reference ID/Investigator# 32125, Toronto, Ontario
  - Site Reference ID/Investigator# 42376, Toronto, Ontario
  - Site Reference ID/Investigator# 32549, Toronto, Ontario
  - Site Reference ID/Investigator# 32540, Toronto, Ontario
  - Site Reference ID/Investigator# 32538, Toronto, Ontario
  - Site Reference ID/Investigator# 37933, Toronto, Ontario
  - Site Reference ID/Investigator# 30874, Toronto, Ontario
  - Site Reference ID/Investigator# 31274, Toronto, Ontario
  - Site Reference ID/Investigator# 37936, Toronto, Ontario
  - Site Reference ID/Investigator# 42436, Toronto, Ontario
  - Site Reference ID/Investigator# 42370, Toronto, Ontario
  - Site Reference ID/Investigator# 30948, Toronto, Ontario
  - Site Reference ID/Investigator# 31336, Toronto, Ontario
  - Site Reference ID/Investigator# 32541, Toronto, Ontario
  - Site Reference ID/Investigator# 37786, Toronto, Ontario
  - Site Reference ID/Investigator# 31295, Toronto, Ontario
  - Site Reference ID/Investigator# 31391, Toronto, Ontario
  - Site Reference ID/Investigator# 37925, Toronto, Ontario
  - Site Reference ID/Investigator# 30953, Toronto, Ontario
  - Site Reference ID/Investigator# 30889, Toronto, Ontario
  - Site Reference ID/Investigator# 30934, Toronto, Ontario
  - Site Reference ID/Investigator# 30869, Toronto, Ontario
  - Site Reference ID/Investigator# 42405, Toronto, Ontario
  - Site Reference ID/Investigator# 42430, Toronto, Ontario
  - Site Reference ID/Investigator# 31377, Toronto, Ontario
  - Site Reference ID/Investigator# 42432, Toronto, Ontario
  - Site Reference ID/Investigator# 32550, Toronto, Ontario
  - Site Reference ID/Investigator# 32547, Toronto, Ontario
  - Site Reference ID/Investigator# 37917, Toronto, Ontario
  - Site Reference ID/Investigator# 42366, Toronto, Ontario
  - Site Reference ID/Investigator# 31378, Toronto, Ontario
  - Site Reference ID/Investigator# 32161, Toronto, Ontario
  - Site Reference ID/Investigator# 47564, Totonto, Ontario
  - Site Reference ID/Investigator# 42372, Waterdown, Ontario
  - Site Reference ID/Investigator# 30902, Welland, Ontario
  - Site Reference ID/Investigator# 32142, Welland, Ontario
  - Site Reference ID/Investigator# 31337, Welland, Ontario
  - Site Reference ID/Investigator# 37883, Whitby, Ontario
  - Site Reference ID/Investigator# 37927, Whitby, Ontario
  - Site Reference ID/Investigator# 37928, Whitby, Ontario
  - Site Reference ID/Investigator# 30931, Whitby, Ontario
  - Site Reference ID/Investigator# 37905, Whitby, Ontario
  - Site Reference ID/Investigator# 37926, Whitby, Ontario
  - Site Reference ID/Investigator# 47577, Whitby, Ontario
  - Site Reference ID/Investigator# 30944, Willowdale, Ontario
  - Site Reference ID/Investigator# 33163, Windsor, Ontario
  - Site Reference ID/Investigator# 37841, Windsor, Ontario
  - Site Reference ID/Investigator# 37776, Windsor, Ontario
  - Site Reference ID/Investigator# 42364, Windsor, Ontario
  - Site Reference ID/Investigator# 30941, Windsor, Ontario
  - Site Reference ID/Investigator# 37738, Windsor, Ontario
  - Site Reference ID/Investigator# 37912, Windsor, Ontario
  - Site Reference ID/Investigator# 30972, Windsor, Ontario
  - Site Reference ID/Investigator# 42346, Windsor, Ontario
  - Site Reference ID/Investigator# 31272, Windsor, Ontario
  - Site Reference ID/Investigator# 42339, Windsor, Ontario
  - Site Reference ID/Investigator# 42456, Windsor, Ontario
  - Site Reference ID/Investigator# 33164, Windsor, Ontario
  - Site Reference ID/Investigator# 31330, Windsor, Ontario
  - Site Reference ID/Investigator# 30875, Windsor, Ontario
  - Site Reference ID/Investigator# 42428, Windsor, Ontario
  - Site Reference ID/Investigator# 42453, Windsor, Ontario
  - Site Reference ID/Investigator# 32150, Windsor, Ontario
  - Site Reference ID/Investigator# 47574, Windsor, Ontario
  - Site Reference ID/Investigator# 42465, Windsor, Ontario
  - Site Reference ID/Investigator# 42371, Woodbridge, Ontario
  - Site Reference ID/Investigator# 31309, Woodbridge, Ontario
  - Site Reference ID/Investigator# 32153, Woodstock, Ontario
  - Site Reference ID/Investigator# 42450, York, Ontario
  - Site Reference ID/Investigator# 33186, York, Ontario
  - Site Reference ID/Investigator# 31273, York, Ontario
  - Site Reference ID/Investigator# 32145, Charlottetown, Prince Edward Island
  - Site Reference ID/Investigator# 32195, Charlottetown, Prince Edward Island
  - Site Reference ID/Investigator# 32221, Charlottetown, Prince Edward Island
  - Site Reference ID/Investigator# 37897, Cornwall, Prince Edward Island
  - Site Reference ID/Investigator# 33019, Kensington, Prince Edward Island
  - Site Reference ID/Investigator# 42470, Summerside, Prince Edward Island
  - Site Reference ID/Investigator# 31267, Alma, Quebec
  - Site Reference ID/Investigator# 37942, Alma, Quebec
  - Site Reference ID/Investigator# 30885, Anjou, Quebec
  - Site Reference ID/Investigator# 31331, Aylmer, Quebec
  - Site Reference ID/Investigator# 31304, Beauceville, Quebec
  - Site Reference ID/Investigator# 31369, Bromont, Quebec
  - Site Reference ID/Investigator# 30903, Brossard, Quebec
  - Site Reference ID/Investigator# 42335, Chicoutimi, Quebec
  - Site Reference ID/Investigator# 31260, Chicoutimi, Quebec
  - Site Reference ID/Investigator# 31398, Clemont, Quebec
  - Site Reference ID/Investigator# 30911, Clermont, Quebec
  - Site Reference ID/Investigator# 31323, Clermont, Quebec
  - Site Reference ID/Investigator# 30928, Cote-St-Luc, Quebec
  - Site Reference ID/Investigator# 42386, Dolbeau-Mistassini, Quebec
  - Site Reference ID/Investigator# 31281, Dolbeau-Mistassini, Quebec
  - Site Reference ID/Investigator# 32182, Gatineau, Quebec
  - Site Reference ID/Investigator# 37937, Gatineau, Quebec
  - Site Reference ID/Investigator# 37843, Gatineau, Quebec
  - Site Reference ID/Investigator# 32910, Gatineau, Quebec
  - Site Reference ID/Investigator# 32911, Gatineau, Quebec
  - Site Reference ID/Investigator# 37941, Gatineau, Quebec
  - Site Reference ID/Investigator# 31393, Grand-Mère, Quebec
  - Site Reference ID/Investigator# 31379, Grand-Mère, Quebec
  - Site Reference ID/Investigator# 37852, Grand-Mère, Quebec
  - Site Reference ID/Investigator# 32141, Grand-Mère, Quebec
  - Site Reference ID/Investigator# 47572, Grande-Allee, Quebec
  - Site Reference ID/Investigator# 30904, Greenfield Park, Quebec
  - Site Reference ID/Investigator# 32966, Hébertville, Quebec
  - Site Reference ID/Investigator# 32167, Hull, Quebec
  - Site Reference ID/Investigator# 31298, Kirkland, Quebec
  - Site Reference ID/Investigator# 32189, L'Anse-Saint-Jean, Quebec
  - Site Reference ID/Investigator# 42344, La Baie, Quebec
  - Site Reference ID/Investigator# 42343, La Malbaie, Quebec
  - Site Reference ID/Investigator# 42377, Lachenaie, Quebec
  - Site Reference ID/Investigator# 30877, Lachute, Quebec
  - Site Reference ID/Investigator# 30968, LaSalle, Quebec
  - Site Reference ID/Investigator# 30918, LaSalle, Quebec
  - Site Reference ID/Investigator# 33042, LaSalle, Quebec
  - Site Reference ID/Investigator# 33046, Laval, Quebec
  - Site Reference ID/Investigator# 31397, Laval, Quebec
  - Site Reference ID/Investigator# 37855, Laval, Quebec
  - Site Reference ID/Investigator# 37856, Laval, Quebec
  - Site Reference ID/Investigator# 42437, Laval, Quebec
  - Site Reference ID/Investigator# 30871, Laval, Quebec
  - Site Reference ID/Investigator# 42402, Laval, Quebec
  - Site Reference ID/Investigator# 31362, Lévis, Quebec
  - Site Reference ID/Investigator# 33062, Lévis, Quebec
  - Site Reference ID/Investigator# 31371, Longueuil, Quebec
  - Site Reference ID/Investigator# 30909, Mistassini, Quebec
  - Site Reference ID/Investigator# 37851, Montreal, Quebec
  - Site Reference ID/Investigator# 31324, Montreal, Quebec
  - Site Reference ID/Investigator# 31308, Montreal, Quebec
  - Site Reference ID/Investigator# 33115, Montreal, Quebec
  - Site Reference ID/Investigator# 42394, Montreal, Quebec
  - Site Reference ID/Investigator# 30921, Montreal, Quebec
  - Site Reference ID/Investigator# 31390, Montreal, Quebec
  - Site Reference ID/Investigator# 33111, Montreal, Quebec
  - Site Reference ID/Investigator# 33110, Montreal, Quebec
  - Site Reference ID/Investigator# 42395, Montreal, Quebec
  - Site Reference ID/Investigator# 30905, Montreal, Quebec
  - Site Reference ID/Investigator# 33112, Montreal, Quebec
  - Site Reference ID/Investigator# 30950, Montreal, Quebec
  - Site Reference ID/Investigator# 31279, Montreal, Quebec
  - Site Reference ID/Investigator# 31293, Montreal, Quebec
  - Site Reference ID/Investigator# 31294, Montreal, Quebec
  - Site Reference ID/Investigator# 33114, Montreal, Quebec
  - Site Reference ID/Investigator# 33116, Montreal, Quebec
  - Site Reference ID/Investigator# 31311, Montreal, Quebec
  - Site Reference ID/Investigator# 32158, Montreal, Quebec
  - Site Reference ID/Investigator#42324, Paspebiac, Quebec
  - Site Reference ID/Investigator# 31372, Plessisville, Quebec
  - Site Reference ID/Investigator# 32133, Plessisville, Quebec
  - Site Reference ID/Investigator# 32437, Plessisville, Quebec
  - Site Reference ID/Investigator# 31370, Pohénégamook, Quebec
  - Site Reference ID/Investigator# 37854, Pointe-aux-Trembles, Quebec
  - Site Reference ID/Investigator# 31332, Pointe-Claire, Quebec
  - Site Reference ID/Investigator# 31358, Pointe-Claire, Quebec
  - Site Reference ID/Investigator# 31392, Princeville, Quebec
  - Site Reference ID/Investigator# 32449, Québec, Quebec
  - Site Reference ID/Investigator# 32159, Québec, Quebec
  - Site Reference ID/Investigator# 32228, Québec, Quebec
  - Site Reference ID/Investigator# 31325, Québec, Quebec
  - Site Reference ID/Investigator# 32603, Québec, Quebec
  - Site Reference ID/Investigator# 32186, Québec, Quebec
  - Site Reference ID/Investigator# 32482, Roxton Pond, Quebec
  - Site Reference ID/Investigator# 31343, Saint Catherine, Quebec
  - Site Reference ID/Investigator# 31283, Saint-Ambroise, Quebec
  - Site Reference ID/Investigator# 31289, Saint-Anselme, Quebec
  - Site Reference ID/Investigator# 31351, Saint-Charles-Borromée, Quebec
  - Site Reference ID/Investigator# 30883, Saint-Henri, Quebec
  - Site Reference ID/Investigator# 31297, Saint-Jérôme, Quebec
  - Site Reference ID/Investigator# 32488, Saint-Lambert-de-Lauzon, Quebec
  - Site Reference ID/Investigator# 32490, Saint-Laurent, Quebec
  - Site Reference ID/Investigator# 32605, Saint-Léonard, Quebec
  - Site Reference ID/Investigator# 32134, Saint-Nicolas, Quebec
  - Site Reference ID/Investigator# 37894, Saint-Pascal, Quebec
  - Site Reference ID/Investigator# 31361, Saint-Pie, Quebec
  - Site Reference ID/Investigator# 37857, Saint-Raymond, Quebec
  - Site Reference ID/Investigator# 32528, Saint-Zacharie, Quebec
  - Site Reference ID/Investigator# 37844, Sainte-Adèle, Quebec
  - Site Reference ID/Investigator# 32135, Sainte-Catherine, Quebec
  - Site Reference ID/Investigator# 32188, Sainte-Claire, Quebec
  - Site Reference ID/Investigator# 31266, Sainte-Julienne, Quebec
  - Site Reference ID/Investigator# 32202, Shefford, Quebec
  - Site Reference ID/Investigator# 31344, Sherbrooke, Quebec
  - Site Reference ID/Investigator# 32509, Sherbrooke, Quebec
  - Site Reference ID/Investigator# 42454, St-Bruno, Quebec
  - Site Reference ID/Investigator# 32526, St-Stanislas-De-Champlain, Quebec
  - Site Reference ID/Investigator# 31341, Ste Felicite, Quebec
  - Site Reference ID/Investigator# 32222, Ste Marie de Beauce, Quebec
  - Site Reference ID/Investigator# 42380, Ste-Marthe-sur-le-Lac, Quebec
  - Site Reference ID/Investigator# 31262, Verdun, Quebec
  - Site Reference ID/Investigator# 30897, Waterville, Quebec
  - Site Reference ID/Investigator# 33157, Westmount, Quebec
  - Site Reference ID/Investigator# 32183, Westmount, Quebec
  - Site Reference ID/Investigator# 37782, Craik, Saskatchewan
  - Site Reference ID/Investigator# 33232, North Battleford, Saskatchewan
  - Site Reference ID/Investigator# 33233, North Battleford, Saskatchewan
  - Site Reference ID/Investigator# 31366, North Battleford, Saskatchewan
  - Site Reference ID/Investigator# 30881, Regina, Saskatchewan
  - Site Reference ID/Investigator# 37726, Regina, Saskatchewan
  - Site Reference ID/Investigator# 32176, Regina, Saskatchewan
  - Site Reference ID/Investigator# 32123, Rosetown, Saskatchewan
  - Site Reference ID/Investigator# 31317, Saskatoon, Saskatchewan
  - Site Reference ID/Investigator# 32179, Saskatoon, Saskatchewan
  - Site Reference ID/Investigator# 32208, Saskatoon, Saskatchewan
  - Site Reference ID/Investigator# 37887, Saskatoon, Saskatchewan
  - Site Reference ID/Investigator# 31292, Saskatoon, Saskatchewan
  - Site Reference ID/Investigator# 32225, Saskatoon, Saskatchewan
  - Site Reference ID/Investigator# 32493, Saskatoon, Saskatchewan
  - Site Reference ID/Investigator# 31387, Saskatoon, Saskatchewan
  - Site Reference ID/Investigator# 30917, Saskatoon, Saskatchewan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 7993 participants were enrolled at 568 study sites in Canada over a period of 24 months.
Pre-assignment Details: Although 3 participants were considered to have violated the protocol because they were not adults (ie, </= 18 years old), they were included in the Intention-to-Treat (ITT) cohort.
Groups:
- All Enrolled Participants (ITT Cohort): Hypertensive participants (diabetics and non-diabetics, with or without isolated systemic hypertension and/or renal dysfunction) who were either naïve to trandolapril or on trandolapril within past 30 days. Trandolapril 0.5, 1.0, 2.0, or 4.0 mg, was prescribed as per usual care. Participants received at least one dose of trandolapril after enrollment.
Period: Overall Study
Arm/Group | All Enrolled Participants (ITT Cohort)
Started | 7993
Participants Conducted Visit 2 (3-month) | 7125
Participants Conducted Visit 3 (6-month) | 5833
Participants Conducted Visit 4(12-month) | 4983
Completed | 4983
Not Completed | 3010
Not completed — Final Status Unknown | 1073
Not completed — Lost to Follow-up | 670
Not completed — Non-serious Adverse Event | 577
Not completed — Withdrawal of Consent | 244
Not completed — Physician Withdrew from Study | 90
Not completed — Non-compliance | 67
Not completed — Blood Pressure Controlled | 49
Not completed — Physician Switched Medication | 26
Not completed — Physician Discontinued Patient | 12
Not completed — Lack of Efficacy | 98
Not completed — Protocol Violation | 75
Not completed — Serious Adverse Event | 27
Not completed — Multiple Reasons | 2

BASELINE CHARACTERISTICS:
Arm/Group | All Enrolled Participants (ITT Cohort)
Number analyzed (Participants) | 7993
Age Continuous [Mean (Standard Deviation); unit: years] | 58.3 (13.1)
Sex/Gender, Customized [Number; unit: participants]
  Female | 3677
  Male | 4283
  Unknown | 33
Region of Enrollment [Number; unit: participants]
  Canada | 7993
Baseline Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min] — Of the participants in the ITT cohort (n=7993), 3965 had eGFR measurements at baseline. Of the diabetic participants in the ITT cohort (n=1883), 1178 had eGFR measurements at baseline.
  mL/min
    All Participants (n=3965) | 76.9 (20.3)
    Diabetic Participants (n=1178) | 77.7 (24.2)
Baseline Microalbuminuria (MAU) [Mean (Standard Deviation); unit: mg/L] — Of the participants in the ITT cohort (n=7993), 2476 had MAU measurements at baseline. Of the diabetic participants in the ITT cohort (n=1883), 1009 had MAU measurements at baseline.
  mg/L
    All Participants (n=2476) | 36.5 (142.2)
    Diabetic Participants (n=1009) | 55.1 (191.5)
Baseline Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mm Hg] — ISH=isolated systolic hypertension. Of the participants in the ITT cohort (n=7993), 7992 had baseline SBP measurements available.
  mm Hg
    All Participants (n=7992) | 150.8 (15.6)
    Diabetic Participants (n=1883) | 145.8 (15.7)
    Renal Dysfunction Participants (n=196) | 147.6 (17.1)
    ISH Participants (n=2207) | 153.0 (10.9)
Baseline Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mm Hg] — Of the participants in the ITT cohort (n=7993), 7991 had baseline DBP measurements available.
  mm Hg
    All Participants (n=7991) | 89.7 (10.7)
    Diabetic Participants (n=1883) | 85.7 (10.5)
    Renal Dysfunction Participants (n=196) | 83.0 (12.0)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Non-Diabetic and Diabetic Participants Meeting Blood Pressure Targets at 3 Months
Description: Blood pressure (BP) targets, as specified in the 2008 CHEP recommendations, were systolic BP (SBP)/diastolic BP (DBP) <140/90 mm Hg for non-diabetic participants, and SBP/DBP <130/80 mm Hg for diabetic participants.
Time Frame: 3 months
Population: Evaluable participants (diabetic and non-diabetic ITT participants with blood pressure measurement at given time point).
Measure: Number; unit: percentage of participants
Groups:
- Non-Diabetic Cohort: The Non-diabetic cohort includes all hypertensive participants who were either naïve to trandolapril or on trandolapril within past 30 days for whom a diagnosis of diabetes was not present at the Baseline visit. Trandolapril 0.5, 1.0, 2.0, or 4.0 mg, was prescribed as per usual care. Participants received at least one dose of trandolapril after enrollment.
- Diabetic Cohort: The Diabetic cohort includes all hypertensive participants who were either naïve to trandolapril or on trandolapril within past 30 days for whom a diagnosis of diabetes was present at the Baseline visit. Trandolapril 0.5, 1.0, 2.0, or 4.0 mg, was prescribed as per usual care. Participants received at least one dose of trandolapril after enrollment.
Arm/Group | Non-Diabetic Cohort | Diabetic Cohort
Number analyzed (Participants) | 5275 | 1605
percentage of participants | 56.0 [54.6 to 57.3] | 28.2 [26.0 to 30.4]

2. Primary Outcome: Percentage of Non-Diabetic and Diabetic Participants Meeting Blood Pressure Targets at 6 Months
Description: as for outcome 1
Time Frame: 6 months
Population: Evaluable participants (diabetic and non-diabetic ITT participants with blood pressure measurement at given time point).
Measure: Number; unit: percentage of participants
Arm/Group | Non-Diabetic Cohort | Diabetic Cohort
Number analyzed (Participants) | 4374 | 1347
percentage of participants | 66.2 [64.8 to 67.6] | 31.1 [28.6 to 33.6]

3. Primary Outcome: Percentage of Non-Diabetic and Diabetic Participants Meeting Blood Pressure Targets at 12 Months
Description: as for outcome 1
Time Frame: 12 months
Population: Evaluable participants (diabetic and non-diabetic ITT participants with blood pressure measurement at given time point).
Measure: Number; unit: percentage of participants
Arm/Group | Non-Diabetic Cohort | Diabetic Cohort
Number analyzed (Participants) | 3751 | 1174
percentage of participants | 72.9 [71.5 to 74.3] | 34.4 [31.7 to 37.1]

4. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) in Blood Pressure (BP)-Controlled and BP-Uncontrolled Diabetics at 3 Months
Description: Diabetics were considered to be "BP-controlled" if BP <130/80 mm Hg. Diabetics were considered to be "BP-uncontrolled" if BP >/=130/80 mm Hg.
Time Frame: Baseline, 3 Months
Population: Evaluable participants (diabetic ITT participants with eGFR measurement at given time point).
Measure: Mean (95% Confidence Interval); unit: mL/min
Groups:
- Diabetic Cohort: BP-Controlled: The Diabetic cohort includes all hypertensive participants who were either naïve to trandolapril or on trandolapril within past 30 days for whom a diagnosis of diabetes was present at the Baseline visit. Trandolapril 0.5, 1.0, 2.0, or 4.0 mg, was prescribed as per usual care. Participants received at least one dose of trandolapril after enrollment. Diabetics were considered to be BP-controlled if BP <130/80 mm Hg.
- Diabetic Cohort: BP-Uncontrolled: The Diabetic cohort includes all hypertensive participants who were either naïve to trandolapril or on trandolapril within past 30 days for whom a diagnosis of diabetes was present at the Baseline visit. Trandolapril 0.5, 1.0, 2.0, or 4.0 mg, was prescribed as per usual care. Participants received at least one dose of trandolapril after enrollment. Diabetics were considered to be BP-uncontrolled if BP >/=130/80 mm Hg.
Arm/Group | Diabetic Cohort | Diabetic Cohort: BP-Controlled | Diabetic Cohort: BP-Uncontrolled
Number analyzed (Participants) | 472 | 153 | 319
mL/min | 0.7 [-2.9 to 4.3] | -1.5 [-3.2 to 0.3] | 1.7 [-3.6 to 7.0]

5. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) in Blood Pressure (BP)-Controlled and BP-Uncontrolled Diabetics at 6 Months
Description: as for outcome 4
Time Frame: Baseline, 6 Months
Population: Evaluable participants (diabetic ITT participants with eGFR measurement at given time point).
Measure: Mean (95% Confidence Interval); unit: mL/min
Arm/Group | Diabetic Cohort | Diabetic Cohort: BP-Controlled | Diabetic Cohort: BP-Uncontrolled
Number analyzed (Participants) | 399 | 133 | 266
mL/min | 0.0 [-1.2 to 1.2] | 0.7 [-1.2 to 2.7] | -0.4 [-1.9 to 1.1]

6. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) in Blood Pressure (BP)-Controlled and BP-Uncontrolled Diabetics at 12 Months
Description: as for outcome 4
Time Frame: Baseline,12 Months
Population: Evaluable participants (diabetic ITT participants with eGFR measurement at given time point).
Measure: Mean (95% Confidence Interval); unit: mL/min
Arm/Group | Diabetic Cohort | Diabetic Cohort: BP-Controlled | Diabetic Cohort: BP-Uncontrolled
Number analyzed (Participants) | 409 | 148 | 261
mL/min | 0.8 [-0.6 to 2.3] | 1.5 [-1.3 to 4.3] | 0.4 [-1.2 to 2.1]

7. Secondary Outcome: Change From Baseline in Microalbuminuria (MAU) at 3 Months
Time Frame: Baseline, 3 Months
Population: Evaluable participants (all participants in the ITT cohort with MAU measurement at given time point).
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | All Enrolled Participants (ITT Cohort)
Number analyzed (Participants) | 764
mg/L | -6.8 [-17.2 to 3.6]

8. Secondary Outcome: Change From Baseline in Microalbuminuria (MAU) at 6 Months
Time Frame: Baseline, 6 Months
Population: Evaluable Participants (all participants in the ITT cohort with MAU measurement at given time point).
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | All Enrolled Participants (ITT Cohort)
Number analyzed (Participants) | 652
mg/L | -5.3 [-16.0 to 5.3]

9. Secondary Outcome: Change From Baseline in Microalbuminuria (MAU) at 12 Months
Time Frame: Baseline, 12 months
Population: Evaluable Participants (all participants in the ITT cohort with MAU measurement at given time point).
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | All Enrolled Participants (ITT Cohort)
Number analyzed (Participants) | 717
mg/L | -6.9 [-15.9 to 2.0]

10. Secondary Outcome: Percentage of Participants With Isolated Systolic Hypertension (ISH) Reaching 2008 CHEP Systolic Blood Pressure (BP) Target After 3 Months of Therapy
Description: The 2008 CHEP systolic BP (SBP) target is <140 mm Hg. Where a participant had an SBP less than the target, the participant's SBP was defined as "controlled."
Time Frame: 3 Months
Population: Evaluable participants (ITT participants with ISH who had blood pressure measurements at given timepoint).
Measure: Number; unit: percentage of participants
Groups:
- Isolated Systolic Hypertension Cohort: The Isolated Systolic Hypertension (ISH) cohort includes all hypertensive participants who were either naïve to trandolapril or on trandolapril within past 30 days who had a baseline systolic blood pressure >/=140 mm Hg and a baseline diastolic blood pressure <90 mm Hg. Trandolapril 0.5, 1.0, 2.0, or 4.0 mg, was prescribed as per usual care. Participants received at least one dose of trandolapril after enrollment.
Arm/Group | Isolated Systolic Hypertension Cohort
Number analyzed (Participants) | 1953
percentage of participants | 58.4 [56.2 to 60.6]

11. Secondary Outcome: Percentage of Participants With Isolated Systolic Hypertension (ISH) Reaching 2008 CHEP Systolic Blood Pressure (BP) Target After 6 Months of Therapy
Description: as for outcome 10
Time Frame: 6 Months
Population: Evaluable participants (ITT participants with ISH who had blood pressure measurements at given timepoint).
Measure: Number; unit: percentage of participants
Arm/Group | Isolated Systolic Hypertension Cohort
Number analyzed (Participants) | 1617
percentage of participants | 67.6 [65.3 to 69.9]

12. Secondary Outcome: Percentage of Participants With Isolated Systolic Hypertension (ISH) Reaching 2008 CHEP Systolic Blood Pressure (BP) Target After 12 Months of Therapy
Description: as for outcome 10
Time Frame: 12 Months
Population: Evaluable participants (ITT participants with ISH who had blood pressure measurements at given timepoint).
Measure: Number; unit: percentage of participants
Arm/Group | Isolated Systolic Hypertension Cohort
Number analyzed (Participants) | 1420
percentage of participants | 74.2 [71.9 to 76.4]

13. Secondary Outcome: Percentage of Participants Reporting Defined Levels of Satisfaction With Current Therapy at Baseline and After 12 Months of Therapy
Description: Satisfaction with therapy at baseline (BL) and 12 months, using a 5-point Likert scale where participants responded to the question "Are you satisfied with your current hypertension therapy?". The range of responses varied from "1 = not at all satisfied" to "5 = extremely satisfied." Responses "2" through "4" were not otherwise defined, but represented increments of more or less satisfaction with current therapy, respectively.
Time Frame: Day 0 (Baseline), 12 months
Population: ITT cohort. n=evaluable participants from the ITT cohort who answered the satisfaction questions at Baseline and 12-Month visits.
Measure: Number; unit: percentage of participants
Arm/Group | All Enrolled Participants (ITT Cohort)
Number analyzed (Participants) | 7993
percentage of participants
  Score=1 at BL (n=7212) | 28.4
  Score=2 at BL (n=7212) | 26.8
  Score=3 at BL (n=7212) | 30.7
  Score=4 at BL (n=7212) | 10.3
  Score=5 at BL (n=7212) | 3.8
  Score=1 at 12 Months (n=4928) | 1.8
  Score=2 at 12 Months (n=4928) | 3.5
  Score=3 at 12 Months (n=4928) | 9.4
  Score=4 at 12 Months (n=4928) | 33.6
  Score=5 at 12 Months (n=4928) | 51.7

14. Other Pre Specified Outcome: Percentage of Participants Achieving 2008 CHEP Targets After 3 Months of Therapy
Description: Blood Pressure (BP) targets, as specified in the 2008 CHEP recommendations, were systolic BP (SBP)/diastolic BP (DBP) <140/90 mm Hg. Where a participant had both an SBP and DBP less than the target, the participant's BP was defined as "controlled."
Time Frame: 3 Months
Population: Evaluable participants (participants in the ITT cohort with blood pressure measurements at given time point).
Measure: Number; unit: percentage of participants
Arm/Group | All Enrolled Participants (ITT Cohort)
Number analyzed (Participants) | 6880
percentage of participants | 58.3 [57.1 to 59.4]

15. Other Pre Specified Outcome: Percentage of Participants Achieving 2008 CHEP Targets After 6 Months of Therapy
Description: as for outcome 14
Time Frame: 6 Months
Population: Evaluable participants (participants in the ITT cohort with blood pressure measurements at given time point).
Measure: Number; unit: percentage of participants
Arm/Group | All Enrolled Participants (ITT Cohort)
Number analyzed (Participants) | 5721
percentage of participants | 68.1 [66.9 to 69.3]

16. Other Pre Specified Outcome: Percentage of Participants Achieving 2008 CHEP Targets After 12 Months of Therapy
Description: as for outcome 14
Time Frame: 12 Months
Population: Evaluable participants (participants in the ITT cohort with blood pressure measurements at given time point).
Measure: Number; unit: percentage of participants
Arm/Group | All Enrolled Participants (ITT Cohort)
Number analyzed (Participants) | 4925
percentage of participants | 74.4 [73.2 to 75.6]

17. Other Pre Specified Outcome: Percentage of Participants With Renal Dysfunction Achieving 2008 CHEP Targets After 3 Months of Therapy
Description: Blood pressure (BP) targets, as specified in the 2008 CHEP recommendations, were systolic BP (SBP)/diastolic BP (DBP) <130/80 mm Hg. Where a participant had both an SBP and DBP less than the target, the participant's BP was defined as "controlled."
Time Frame: 3 Months
Population: Evaluable participants (ITT participants with renal dysfunction who had blood pressure measurements at given timepoint).
Measure: Number; unit: percentage of participants
Groups:
- Renal Dysfunction Cohort: The Renal Dysfunction cohort includes all hypertensive participants who were either naïve to trandolapril or on trandolapril within past 30 days for whom a co-morbidity of "renal dysfunction" was recorded at the Baseline visit. Trandolapril 0.5, 1.0, 2.0, or 4.0 mg, was prescribed as per usual care. Participants received at least one dose of trandolapril after enrollment.
Arm/Group | Renal Dysfunction Cohort
Number analyzed (Participants) | 172
percentage of participants | 29.1 [22.3 to 35.9]

18. Other Pre Specified Outcome: Percentage of Participants With Renal Dysfunction Achieving 2008 CHEP Targets After 6 Months of Therapy
Description: as for outcome 17
Time Frame: 6 Months
Population: Evaluable participants (ITT participants with renal dysfunction who had blood pressure measurements at given timepoint).
Measure: Number; unit: percentage of participants
Arm/Group | Renal Dysfunction Cohort
Number analyzed (Participants) | 131
percentage of participants | 31.3 [23.4 to 39.2]

19. Other Pre Specified Outcome: Percentage of Participants With Renal Dysfunction Achieving 2008 CHEP Targets After 12 Months of Therapy
Description: as for outcome 17
Time Frame: 12 Months
Population: Evaluable participants (ITT participants with renal dysfunction who had blood pressure measurements at given timepoint).
Measure: Number; unit: percentage of participants
Arm/Group | Renal Dysfunction Cohort
Number analyzed (Participants) | 112
percentage of participants | 36.6 [27.7 to 45.5]

20. Other Pre Specified Outcome: Mean Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) in ITT Cohort at 3 Months
Time Frame: Day 0 (Baseline), 3 Months
Population: ITT cohort. n = all evaluable participants in the ITT cohort with blood pressure measurement at given timepoint.
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | All Enrolled Participants (ITT Cohort)
Number analyzed (Participants) | 7993
mm Hg
  SBP (n=6881) | -16.5 [-16.9 to -16.1]
  DBP (n=6880) | -8.4 [-8.7 to -8.2]

21. Other Pre Specified Outcome: Mean Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) in ITT Cohort at 6 Months
Time Frame: Day 0 (Baseline), 6 Months
Population: Evaluable participants (participants in the ITT cohort with blood pressure measurements at given time point).
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | All Enrolled Participants (ITT Cohort)
Number analyzed (Participants) | 5721
mm Hg
  SBP | -18.7 [-19.2 to -18.3]
  DBP | -9.7 [-10.8 to -9.4]

22. Other Pre Specified Outcome: Mean Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) in ITT Cohort at 12 Months
Time Frame: Day 0 (Baseline), 12 Months
Population: Evaluable participants (participants in the ITT cohort with blood pressure measurements at given timepoint).
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | All Enrolled Participants (ITT Cohort)
Number analyzed (Participants) | 4925
mm Hg
  SBP | -20.1 [-20.6 to -19.6]
  DBP | -10.5 [-10.8 to -10.2]

23. Other Pre Specified Outcome: Mean Baseline Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) in Non-Diabetic, Diabetic, ISH, and Renal Dysfunction Cohorts
Time Frame: Day 0 (Baseline)
Population: Evaluable participants (ITT participants in the non-diabetic, diabetic, ISH, and renal dysfunction cohorts with blood pressure measurement at timepoint).
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Non-Diabetic Cohort | Diabetic Cohort | Isolated Systolic Hypertension Cohort | Renal Dysfunction Cohort
Number analyzed (Participants) | 6108 | 1883 | 2207 | 196
mm Hg
  SBP | 152.4 [152.0 to 152.8] | 145.8 [145.1 to 146.5] | 153.3 [152.9 to 153.8] | 147.6 [145.2 to 150]
  DBP | 90.9 [90.7 to 91.2] | 85.7 [85.2 to 86.1] | 80.2 [79.9 to 80.4] | 83.0 [81.3 to 84.7]

24. Other Pre Specified Outcome: Mean Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) in Non-Diabetic, Diabetic, ISH, and Renal Dysfunction Cohorts at Month 3
Time Frame: Day 0 (Baseline), Month 3
Population: as for outcome 23
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Non-Diabetic Cohort | Diabetic Cohort | Isolated Systolic Hypertension Cohort | Renal Dysfunction Cohort
Number analyzed (Participants) | 5275 | 1605 | 1953 | 172
mm Hg
  SBP | -17.4 [-17.8 to -16.9] | -13.6 [-14.4 to -12.8] | -17.2 [-17.9 to -16.5] | -14.8 [-17.6 to -12.1]
  DBP | -8.8 [-9.1 to -8.5] | -7.0 [-7.5 to -6.5] | -2.5 [-2.9 to -2.1] | -6.9 [-8.7 to -5.2]

25. Other Pre Specified Outcome: Mean Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) in Non-Diabetic, Diabetic, ISH, and Renal Dysfunction Cohorts at Month 6
Time Frame: Day 0 (Baseline), Month 6
Population: as for outcome 23
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Non-Diabetic Cohort | Diabetic Cohort | Isolated Systolic Hypertension Cohort | Renal Dysfunction Cohort
Number analyzed (Participants) | 4374 | 1347 | 1617 | 131
mm Hg
  SBP | -19.8 [-20.3 to -19.3] | -15.3 [-16.1 to -14.4] | -19.2 [-19.9 to -18.4] | -17.5 [-20.6 to -14.3]
  DBP | -10.3 [-10.6 to -9.9] | -7.9 [-8.4 to -7.3] | -2.9 [-3.4 to -2.5] | -8.2 [-10.2 to -6.1]

26. Other Pre Specified Outcome: Mean Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) in Non-Diabetic, Diabetic, ISH, and Renal Dysfunction Cohorts at Month 12
Time Frame: Day 0 (Baseline), Month 12
Population: as for outcome 23
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Non-Diabetic Cohort | Diabetic Cohort | Isolated Systolic Hypertension Cohort | Renal Dysfunction Cohort
Number analyzed (Participants) | 3751 | 1174 | 1420 | 112
mm Hg
  SBP | -21.2 [-21.7 to -20.6] | -16.7 [-17.6 to -15.7] | -20.5 [-21.2 to -19.7] | -18.3 [-21.8 to -14.8]
  DBP | -11.0 [-11.4 to -10.7] | -8.8 [-9.4 to -8.2] | -3.6 [-4.0 to -3.1] | -9.7 [-11.8 to -7.6]

27. Other Pre Specified Outcome: Number of Participants Compliant With Therapy After 3 Months
Description: Compliance after 3 months of treatment was derived using responses to the Visit 2 question "How many trandolapril (Mavik®) doses have been missed since the subject's last visit?" If the response was "zero", the participant was classified as "compliant." If the response was any value greater than zero, regardless of the number of missed doses, the participant was classified as "non-compliant."
Time Frame: 3 Months
Population: Evaluable participants (participants in the ITT cohort with compliance data available at given time point).
Measure: Number; unit: participants
Arm/Group | All Enrolled Participants (ITT Cohort)
Number analyzed (Participants) | 6716
participants | 5015 [73.6 to 75.7]

28. Other Pre Specified Outcome: Number of Participants Compliant With Therapy After 6 Months
Description: Compliance after 6 months of treatment was derived using responses to the question "How many trandolapril (Mavik®) doses have been missed since the subject's last visit?" at both Visit 2 and Visit 3, as follows: If the response was "zero" at both the Visit 2 and Visit 3 assessments, participant was classified as "compliant" after 6 months of treatment; If the response was any value greater than zero at either of the Visit 2 or Visit 3 assessments, regardless of the number of missed doses, participant was classified as "non-compliant" after 6 months of treatment
Time Frame: 6 Months
Population: Evaluable participants (participants in the ITT cohort with compliance data available at given time point).
Measure: Number; unit: participants
Arm/Group | All Enrolled Participants (ITT Cohort)
Number analyzed (Participants) | 5588
participants | 3661 [64.3 to 66.8]

29. Other Pre Specified Outcome: Number of Participants Compliant With Therapy After 12 Months
Description: Compliance after 12 months of treatment was derived using responses to the question "How many trandolapril doses have been missed since the subject's last visit?" at Visit 2, Visit 3 and Visit 4, as follows: if the response was "zero" at all of the Visits 2 through 4 assessments, the participant was classified as "compliant" after 12 months of treatment; if the response was any value greater than zero at any of the Visits 2 through 4 assessments, regardless of the number of missed doses, the participant was classified as "non-compliant" after 12 months of treatment.
Time Frame: 12 Months
Population: Evaluable participants (participants in the ITT cohort with compliance data available at given time point).
Measure: Number; unit: participants
Arm/Group | All Enrolled Participants (ITT Cohort)
Number analyzed (Participants) | 4728
participants | 2793 [57.7 to 60.5]

30. Other Pre Specified Outcome: Number of Participants With Dose Changes at 3 Months
Time Frame: 3 Months
Population: Evaluable participants (all participants in the ITT cohort with data available at given time point).
Measure: Number; unit: participants
Arm/Group | All Enrolled Participants (ITT Cohort)
Number analyzed (Participants) | 6456
participants
  Dose Decreased | 173
  Dose Increased | 1868
  No Change in Dose | 4373
  Unknown | 42

31. Other Pre Specified Outcome: Number of Participants With Dose Changes at 6 Months
Time Frame: 6 Months
Population: Evaluable participants (all participants in the ITT cohort with data available at given time point).
Measure: Number; unit: participants
Arm/Group | All Enrolled Participants (ITT Cohort)
Number analyzed (Participants) | 5519
participants
  Dose Decreased | 125
  Dose Increased | 578
  No Change in Dose | 4735
  Unknown | 81

32. Other Pre Specified Outcome: Number of Participants With Dose Changes at 12 Months
Time Frame: 12 Months
Population: Evaluable participants (all participants in the ITT cohort with data available at given time point).
Measure: Number; unit: participants
Arm/Group | All Enrolled Participants (ITT Cohort)
Number analyzed (Participants) | 4770
participants
  Dose Decreased | 100
  Dose Increased | 370
  No Change in Dose | 4196
  Unknown | 104

33. Other Pre Specified Outcome: Percentage of Diabetic and Non-diabetic (Blood Pressure [BP]-Controlled and BP-Uncontrolled) Participants With Dose Increases After 3 Months
Description: The percentage of non-diabetic and diabetic participants whose systolic and diastolic blood pressures were "controlled" versus "uncontrolled" was assessed using 2008 CHEP-specified targets (non-diabetics: BP <140/90 mm Hg; diabetics: BP <130/80 mm Hg). The percentage of these "controlled" and "uncontrolled" participants who underwent or did not undergo a dose increase is presented.
Time Frame: 3 Months
Population: Evaluable participants (diabetic and non-diabetic ITT participants with available data at given time point).
Measure: Number; unit: percentage of participants
Groups:
- Non-Diabetic Cohort: BP-Uncontrolled: The Non-diabetic cohort includes all hypertensive participants who were either naïve to trandolapril or on trandolapril within past 30 days for whom a diagnosis of diabetes was not present at the Baseline visit. Trandolapril 0.5, 1.0, 2.0, or 4.0 mg, was prescribed as per usual care. Participants received at least one dose of trandolapril after enrollment. Non-diabetics were considered to be BP-uncontrolled if BP >/=140/90 mm Hg.
- Non-Diabetic Cohort: BP-Controlled: The Non-diabetic cohort includes all hypertensive participants who were either naïve to trandolapril or on trandolapril within past 30 days for whom a diagnosis of diabetes was not present at the Baseline visit. Trandolapril 0.5, 1.0, 2.0, or 4.0 mg, was prescribed as per usual care. Participants received at least one dose of trandolapril after enrollment. Non-diabetics were considered to be BP-controlled if BP <140/90 mm Hg.
Arm/Group | Non-Diabetic Cohort: BP-Uncontrolled | Non-Diabetic Cohort: BP-Controlled | Diabetic Cohort: BP-Uncontrolled | Diabetic Cohort: BP-Controlled
Number analyzed (Participants) | 2115 | 2760 | 1077 | 413
percentage of participants
  Dose Increase | 46.7 | 17.9 | 31.4 | 10.4
  No Dose Increase | 53.3 | 82.1 | 68.6 | 89.6

34. Other Pre Specified Outcome: Percentage of Diabetic and Non-diabetic (Blood Pressure [BP]-Controlled and BP-Uncontrolled) Participants With Dose Increases After 6 Months
Description: as for outcome 33
Time Frame: 6 Months
Population: Evaluable participants (diabetic and non-diabetic ITT participants with available data at given time point).
Measure: Number; unit: percentage of participants
Arm/Group | Non-Diabetic Cohort: BP-Uncontrolled | Non-Diabetic Cohort: BP-Controlled | Diabetic Cohort: BP-Uncontrolled | Diabetic Cohort: BP-Controlled
Number analyzed (Participants) | 1357 | 2785 | 870 | 406
percentage of participants
  Dose Increase | 23.1 | 4.9 | 12.1 | 5.4
  No Dose Increase | 76.9 | 95.1 | 87.9 | 94.6

35. Other Pre Specified Outcome: Percentage of Diabetic and Non-diabetic (Blood Pressure [BP]-Controlled and BP-Uncontrolled) Participants With Dose Increases After 12 Months
Description: as for outcome 33
Time Frame: 12 Months
Population: Evaluable participants (diabetic and non-diabetic ITT participants with available data at given time point).
Measure: Number; unit: percentage of participants
Arm/Group | Non-Diabetic Cohort: BP-Uncontrolled | Non-Diabetic Cohort: BP-Controlled | Diabetic Cohort: BP-Uncontrolled | Diabetic Cohort: BP-Controlled
Number analyzed (Participants) | 912 | 2630 | 712 | 393
percentage of participants
  Dose Increase | 15.7 | 5.2 | 9.6 | 4.8
  No Dose Increase | 84.3 | 94.8 | 90.4 | 95.2

36. Other Pre Specified Outcome: Number of Participants Adding Concomitant Cardiovascular Medications at 3 Months
Description: Presented by type of medication added.
Time Frame: 3 Months
Population: Evaluable participants (all participants in the ITT cohort with available data at given time point).
Measure: Number; unit: participants
Arm/Group | All Enrolled Participants (ITT Cohort)
Number analyzed (Participants) | 7125
participants
  None | 6090
  Diuretic | 284
  Angiotensin receptor blocker | 133
  Calcium channel blocker | 186
  Beta-blocker | 78

37. Other Pre Specified Outcome: Number of Participants Adding Concomitant Cardiovascular Medications at 6 Months
Description: Presented by type of medication added.
Time Frame: 6 Months
Population: Evaluable participants (all participants in the ITT cohort with available data at given time point).
Measure: Number; unit: participants
Arm/Group | All Enrolled Participants (ITT Cohort)
Number analyzed (Participants) | 5833
participants
  None | 5193
  Diuretic | 222
  Angiotensin receptor blocker | 82
  Calcium channel blocker | 123
  Beta-blocker | 41

38. Other Pre Specified Outcome: Number of Participants Adding Concomitant Cardiovascular Medications at 12 Months
Description: Presented by type of medication added.
Time Frame: 12 Months
Population: Evaluable participants (all participants in the ITT cohort with available data at given time point).
Measure: Number; unit: participants
Arm/Group | All Enrolled Participants (ITT Cohort)
Number analyzed (Participants) | 4983
participants
  None | 4540
  Diuretic | 144
  Angiotensin receptor blocker | 61
  Calcium channel blocker | 86
  Beta-blocker | 35

39. Other Pre Specified Outcome: Number of Participants Discontinuing Concomitant Cardiovascular Medications at 3 Months
Description: Presented by type of medication discontinued.
Time Frame: 3 Months
Population: Evaluable participants (all participants in the ITT cohort with available data at given time point).
Measure: Number; unit: participants
Arm/Group | All Enrolled Participants (ITT Cohort)
Number analyzed (Participants) | 7125
participants
  None | 6656
  Diuretic | 27
  Angiotensin-converting-enzyme inhibitor | 4
  Angiotensin receptor blocker | 6
  Calcium channel blocker | 22
  Beta-blocker | 20

40. Other Pre Specified Outcome: Number of Participants Discontinuing Concomitant Cardiovascular Medications at 6 Months
Description: Presented by type of medication discontinued.
Time Frame: 6 Months
Population: Evaluable participants (all participants in the ITT cohort with available data at given time point).
Measure: Number; unit: participants
Arm/Group | All Enrolled Participants (ITT Cohort)
Number analyzed (Participants) | 5833
participants
  None | 5607
  Diuretic | 24
  Angiotensin-converting-enzyme inhibitor | 4
  Angiotensin receptor blocker | 4
  Calcium channel blocker | 17
  Beta-blocker | 8

41. Other Pre Specified Outcome: Number of Participants Discontinuing Concomitant Cardiovascular Medications at 12 Months
Description: Presented by type of medication discontinued.
Time Frame: 12 Months
Population: Evaluable participants (all participants in the ITT cohort with available data at given time point).
Measure: Number; unit: participants
Arm/Group | All Enrolled Participants (ITT Cohort)
Number analyzed (Participants) | 4983
participants
  None | 4823
  Diuretic | 25
  Angiotensin-converting-enzyme inhibitor | 2
  Angiotensin receptor blocker | 3
  Calcium channel blocker | 10
  Beta-blocker | 6

42. Other Pre Specified Outcome: Percentage of Diabetic and Renal Dysfunction Participants Achieving the Target of Blood Pressure (BP) <140/90 mm Hg at 3 Months
Description: Participants achieving the target of blood pressure <140/90 mm Hg were considered "controlled."
Time Frame: 3 Months
Population: Evaluable participants (ITT participants in the Diabetic or Renal Dysfunction cohorts with BP measurement at given time point).
Measure: Number; unit: percentage of participants
Arm/Group | Diabetic Cohort | Renal Dysfunction Cohort
Number analyzed (Participants) | 1605 | 172
percentage of participants | 65.7 [63.4 to 68.0] | 66.3 [59.2 to 73.3]

43. Other Pre Specified Outcome: Percentage of Diabetic and Renal Dysfunction Participants Achieving the Target of Blood Pressure (BP) <140/90 mm Hg at 6 Months
Description: Participants achieving the target of blood pressure <140/90 mm Hg were considered "controlled."
Time Frame: 6 Months
Population: Evaluable participants (ITT participants in the Diabetic or Renal Dysfunction cohorts with blood pressure measurement at given time point).
Measure: Number; unit: percentage of participants
Arm/Group | Diabetic Cohort | Renal Dysfunction Cohort
Number analyzed (Participants) | 1347 | 131
percentage of participants | 74.1 [71.8 to 76.4] | 70.2 [62.4 to 78.1]

44. Other Pre Specified Outcome: Percentage of Diabetic and Renal Dysfunction Participants Achieving the Target of Blood Pressure (BP) <140/90 mm Hg at 12 Months
Description: Participants achieving the target of blood pressure <140/90 mm Hg were considered "controlled."
Time Frame: 12 Months
Population: as for outcome 42
Measure: Number; unit: percentage of participants
Arm/Group | Diabetic Cohort | Renal Dysfunction Cohort
Number analyzed (Participants) | 1174 | 112
percentage of participants | 79.2 [76.9 to 81.5] | 75.0 [67.0 to 83.0]

45. Secondary Outcome: Percentage of Participants Reporting Defined Levels of Satisfaction With Current Therapy at Baseline Versus After 12 Months of Therapy
Description: Satisfaction with therapy at baseline (BL) versus 12 months, using a 5-point Likert scale where participants responded to the question "Are you satisfied with your current hypertension therapy?". The range of responses varied from "1 = not at all satisfied" to "5 = extremely satisfied." Responses "2" through "4" were not otherwise defined, but represented increments of more or less satisfaction with current therapy, respectively.
Time Frame: Day 0 (Baseline), 12 months
Population: Subset of participants from the ITT cohort who answered the satisfaction questions at both the Baseline and 12-Month visits.
Measure: Number; unit: percentage of participants
Arm/Group | All Enrolled Participants (ITT Cohort)
Number analyzed (Participants) | 4510
percentage of participants
  Score=1 (at BL) / Score=1 (at 12 Months) | 0.62
  Score=1 (at BL) / Score=2 (at 12 Months) | 0.67
  Score=1 (at BL) / Score=3 (at 12 Months) | 2.33
  Score=1 (at BL) / Score=4 (at 12 Months) | 8.36
  Score=1 (at BL) / Score=5 (at 12 Months) | 15.63
  Score=2 (at BL) / Score=1 (at 12 Months) | 0.42
  Score=2 (at BL) / Score=2 (at 12 Months) | 1.82
  Score=2 (at BL) / Score=3 (at 12 Months) | 2.71
  Score=2 (at BL) / Score=4 (at 12 Months) | 9.84
  Score=2 (at BL) / Score=5 (at 12 Months) | 11.82
  Score=3 (at BL) / Score=1 (at 12 Months) | 0.53
  Score=3 (at BL) / Score=2 (at 12 Months) | 0.89
  Score=3 (at BL) / Score=3 (at 12 Months) | 3.90
  Score=3 (at BL) / Score=4 (at 12 Months) | 12.06
  Score=3 (at BL) / Score=5 (at 12 Months) | 13.86
  Score=4 (at BL) / Score=1 (at 12 Months) | 0.07
  Score=4 (at BL) / Score=2 (at 12 Months) | 0.09
  Score=4 (at BL) / Score=3 (at 12 Months) | 0.53
  Score=4 (at BL) / Score=4 (at 12 Months) | 4.12
  Score=4 (at BL) / Score=5 (at 12 Months) | 5.96
  Score=5 (at BL) / Score=1 (at 12 Months) | 0.07
  Score=5 (at BL) / Score=2 (at 12 Months) | 0.07
  Score=5 (at BL) / Score=3 (at 12 Months) | 0.29
  Score=5 (at BL) / Score=4 (at 12 Months) | 0.67
  Score=5 (at BL) / Score=5 (at 12 Months) | 2.68

ADVERSE EVENTS:
Time Frame: Day 0 to Day 360
Arm/Group | All Enrolled Participants (ITT Cohort)
Serious Adverse Events (participants affected / at risk) | 83/7993
Other Adverse Events (participants affected / at risk) | 527/7993
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Enrolled Participants (ITT Cohort) (N=7993)
pneumonia (Infections and infestations) | 3
sepsis (Infections and infestations) | 3
gangrene (Infections and infestations) | 1
lung infection (Infections and infestations) | 1
lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
amyloidosis (Immune system disorders) | 1
hypothyroidism (Endocrine disorders) | 1
diabetes mellitus (Metabolism and nutrition disorders) | 2
hyponatraemia (Metabolism and nutrition disorders) | 1
alcoholism (Psychiatric disorders) | 1
completed suicide (Psychiatric disorders) | 1
schizophrenia (Psychiatric disorders) | 1
cerebrovascular accident (Nervous system disorders) | 5
dizziness (Nervous system disorders) | 3
syncope (Nervous system disorders) | 1
carotid artery stenosis (Nervous system disorders) | 1
cerebral hematoma (Nervous system disorders) | 1
coma (Nervous system disorders) | 1
dementia (Nervous system disorders) | 1
loss of consciousness (Nervous system disorders) | 1
quadriplegia (Nervous system disorders) | 1
transient ischemic attack (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
eye haemorrhage (Eye disorders) | 1
ocular vascular disorder (Eye disorders) | 1
visual acuity reduced (Eye disorders) | 1
myocardial infarction (Cardiac disorders) | 8
atrial fibrillation (Cardiac disorders) | 5
angina pectoris (Cardiac disorders) | 4
cardiac arrest (Cardiac disorders) | 3
cardiac failure (Cardiac disorders) | 3
cardiac failure congestive (Cardiac disorders) | 3
acute coronary syndrome (Cardiac disorders) | 2
cardiac disorder (Cardiac disorders) | 2
coronary artery disease (Cardiac disorders) | 2
coronary artery stenosis (Cardiac disorders) | 2
palpitations (Cardiac disorders) | 2
ventricular hypokinesis (Cardiac disorders) | 1
arteriosclerosis coronary artery (Cardiac disorders) | 1
atrioventricular block (Cardiac disorders) | 1
bradycardia (Cardiac disorders) | 1
cardiac tamponade (Cardiac disorders) | 1
cardiogenic shock (Cardiac disorders) | 1
cardio-respiratory arrest (Cardiac disorders) | 1
coronary artery occlusion (Cardiac disorders) | 1
coronary artery thrombosis (Cardiac disorders) | 1
left ventricular dysfunction (Cardiac disorders) | 1
left ventricular hypertrophy (Cardiac disorders) | 1
mitral valve disease (Cardiac disorders) | 1
mitral valve incompetence (Cardiac disorders) | 1
myocardial ischemia (Cardiac disorders) | 1
pericardial haemorrhage (Cardiac disorders) | 1
right ventricular dysfunction (Cardiac disorders) | 1
sick sinus syndrome (Cardiac disorders) | 1
supraventricular tachycardia (Cardiac disorders) | 1
torsade de pointes (Cardiac disorders) | 1
ventricular fibrillation (Cardiac disorders) | 1
infarction (Vascular disorders) | 2
aortic aneurysm (Vascular disorders) | 1
arterial occlusive disease (Vascular disorders) | 1
arteriosclerosis (Vascular disorders) | 1
blood pressure inadequately controlled (Vascular disorders) | 1
hypotension (Vascular disorders) | 1
peripheral ischaemia (Vascular disorders) | 1
peripheral vascular disease (Vascular disorders) | 1
shock (Vascular disorders) | 1
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
pulmonary oedema (Vascular disorders) | 3
cough (Respiratory, thoracic and mediastinal disorders) | 2
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
abdominal pain (Gastrointestinal disorders) | 2
pancreatitis acute (Gastrointestinal disorders) | 2
ascites (Gastrointestinal disorders) | 1
colitis iscaemic (Gastrointestinal disorders) | 1
gastric ulcer (Gastrointestinal disorders) | 1
gastroesophageal reflux disease (Gastrointestinal disorders) | 1
hiatus hernia (Gastrointestinal disorders) | 1
lip swelling (Gastrointestinal disorders) | 1
oedema mouth (Gastrointestinal disorders) | 1
swollen tongue (Gastrointestinal disorders) | 1
angioedema (Skin and subcutaneous tissue disorders) | 1
pain in extremity (Musculoskeletal and connective tissue disorders) | 2
lower extremity mass (Musculoskeletal and connective tissue disorders) | 1
mobility decreased (Musculoskeletal and connective tissue disorders) | 1
renal failure (Renal and urinary disorders) | 2
glomerulonephritis membranous (Renal and urinary disorders) | 1
oliguria (Renal and urinary disorders) | 1
proteinuria (Renal and urinary disorders) | 1
renal failure acute (Renal and urinary disorders) | 1
post-menopausal haemorrhage (Reproductive system and breast disorders) | 1
death (General disorders) | 5
chest pain (General disorders) | 4
asthenia (General disorders) | 3
fatigue (General disorders) | 2
oedema peripheral (General disorders) | 2
chest discomfort (General disorders) | 1
malaise (General disorders) | 1
terminal state (General disorders) | 1
weight decreased (Investigations) | 2
blood pressure decreased (Investigations) | 1
fall (Injury, poisoning and procedural complications) | 4
hip fracture (Injury, poisoning and procedural complications) | 2
post-procedural complication (Injury, poisoning and procedural complications) | 2
road traffic accident (Injury, poisoning and procedural complications) | 2
complications of transplanted liver (Injury, poisoning and procedural complications) | 1
femur fracture (Injury, poisoning and procedural complications) | 1
foot fracture (Injury, poisoning and procedural complications) | 1
injury (Injury, poisoning and procedural complications) | 1
lower limb fracture (Injury, poisoning and procedural complications) | 1
rib fracture (Injury, poisoning and procedural complications) | 1
pericardial drainage (Surgical and medical procedures) | 1
aortic valve replacement (Surgical and medical procedures) | 1
cardiac pacemaker insertion (Surgical and medical procedures) | 1
hernia hiatus repair (Surgical and medical procedures) | 1
hospitalization (Surgical and medical procedures) | 1
knee arthroplasty (Surgical and medical procedures) | 1
rotator cuff repair (Surgical and medical procedures) | 1
homicide (Social circumstances) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Enrolled Participants (ITT Cohort) (N=7993)
cough (Respiratory, thoracic and mediastinal disorders) | 527 — Cough is an expected event for this class of drugs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.